CLINICAL TRIAL: NCT03723798
Title: A Multicenter, Placebo Controlled, 4-group Parallel Randomized, Double Blind, Phase II Study to Evaluate the Efficacy and Safety of Orally Administered SA001 in Patients With Dry Eye Syndrome.
Brief Title: Clinical Study to Investigate the Efficacy and Safety of Orally Administered SA001 in Patients With Dry Eye Syndrome.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samjin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SJSA001_03
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): SA001 Low dose
  Interventions: Drug: SA001 Low dose
- Group 2 (Experimental): SA001 Mid dose
  Interventions: Drug: SA001 Mid dose
- Group 3 (Experimental): SA001 High dose
  Interventions: Drug: SA001 High dose
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SA001 Low dose — 3 tablets b.i.d for 12 weeks
  Arms: Group 1
Drug: SA001 Mid dose — 3 tablets b.i.d for 12 weeks
  Arms: Group 2
Drug: SA001 High dose — 3 tablets b.i.d for 12 weeks
  Arms: Group 3
Drug: Placebo — 3 tablets b.i.d for 12 weeks
  Arms: Placebo

SUMMARY:
This is a phase 2, multicenter, double-blind, placebo control, randomized study to evaluate the efficacy and safety of orally administered SA001 compared to placebo in patients with Dry Eye Syndrome.

The clinical trial consists of a wash-out period of 14 days, a treatment period of 12 weeks, and a follow-up period of 1 week after administration of the Investigational Product. If the subject voluntarily signs the informed consent form(ICF), the investigator conducts screening tests and check medical history to evaluate the subject's suitability. As a result of the screening test, eligible subjects should stop using the prior medication for dry eye syndrome during the 14 days of observation period, and if necessary, subjects can use rescue drug(artificial tears) for the first 11 days, and then discontinue all eye drops including rescue drug(artificial tears) for 3 days. And all of these subjects will be randomized in a 1:1:1:1 ratio to receive 3 different doses of investigational product (SA001 or placebo) everyday for 12 weeks. During the treatment period, If necessary, subjects can use the rescue drug (artificial tears), and the number of administration of rescue drug is limited to 3 times a day, and when used, the administration time should be recorded in the subject's diary.

Subjects should visit to the study site on 2, 4, 8 and 12 weeks after starting dosing investigational product. Efficacy evaluation results are collected from both eyes, and the primary evaluation variable is analyzed using the test results collected from 'Worse eye' (the eye with the worse keratoconjunctival staining result among both eyes). Worse eye will be determined at the baseline visit and, if the results of both eyes are the same, the test result of the left eye is used.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 19
2. Patient who meets all of the following criteria in at least one of both eyes

   * Fluorescein corneal staining score ≥ 2
   * Schirmer test ≤ 10mm in 5 mins
   * Tear break-up time ≤ 10 secs
3. Patient who diagnosed with dry eye syndrome at the time of screening and who have dry eye symptoms (dryness, discomfort, foreign body sensation, pain, vision fluctuation, etc.)
4. Patient who agrees not to use eye drops other than the rescue drugs provided during the clinical trial period
5. Patient who can understand the clinical trial and voluntarily signs an informed consent

Exclusion Criteria:

1. Clinically significant ophthalmic diseases not caused by dry eye disease (corneal surface disease, abnormal corneal sensitivity, abnormal tear excess, etc.) that may confuse the interpretation of clinical trial results
2. In case of being treated with anti-inflammatory therapy for dry eye, such as steroid or non-steroidal anti-inflammatory eye drops, autologous serum eye drops, etc.
3. In case of administration of steroids or immunosuppressants (azathioprine, tacrolimus, cyclosporine, mofetil mycophenolate, etc.)
4. Patient who has worn contact lenses within 72 hours prior to screening or need to wear contact lenses during the clinical trial period
5. A history of intraocular surgery within 90 days prior to screening
6. Active eye infection symptoms such as anterior uveitis, anterior blepharitis, and Steven-Johnson syndrome
7. Patient with an eye allergy or who are currently receiving treatment for an allergic eye disease (using antihistamines, etc.)
8. Autoimmune disease (ex. Sjögren's syndrome, Rheumatoid arthritis, systemic lupus erythematosus, Graves' disease, etc.)
9. Patient who needs surgery due to surface elevation caused by Meibomian Gland Dysfunction (MGD)
10. A history of corneal transplantation or neurotrophic keratitis
11. Patient who has an intraocular pressure of 25 mmHg or higher in one or more of both eyes or have been diagnosed with glaucoma
12. Patient who has undergone vision correction surgery such as LASIK (Laser-Assisted in Situ Keratomileusis) within 12 months prior to screening
13. Patient who has undergone silicone lacrimal punctal occlusion or cauterization of the punctum within 90 days prior to screening. However, patient who has undergone collagen lacrimal punctal occlusion can be enrolled.
14. Hypersensitivity to the ingredients of the investigational product including rebamipide
15. Clinically significant liver, kidney, nervous system, immune system, respiratory or endocrine disease, blood/tumor disease, cardiovascular disease, mental disease (mood disorder, obsessive-compulsive disorder, etc.) or a history of those diseases
16. Patient who shows the following examination findings at visit 1 (screening visit)

    * WBC ≤ 4,000/mm3
    * Platelets ≤ 100,000/mm3
    * AST/ALT/ALP ≥ 3 times the upper limit of normal(ULN)
    * Total bilirubin ≥ 1.5 times the upper limit of normal(ULN)
17. A woman who has a positive Serum hCG test at the screening visit (Visit 1), or who does not agree to use at least one effective contraceptive method that is medically acceptable
18. Take oral contraceptives during the study period
19. Pregnant or lactating women
20. A history of drug or alcohol abuse
21. Participation in an investigational drug or device trial within 30 days prior to screening
22. Any condition that, in the opinion of the investigator, would inappropriate to participate in the clinical trial

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-08 (Actual)

PRIMARY OUTCOMES:
Change in Fluorescein Corneal Staining(FCS) score from baseline to Day 84 | Baseline(Day0) and Day 84

SECONDARY OUTCOMES:
Change in Fluorescein Corneal Staining(FCS) score from baseline to Day 14, Day 28 and Day 56 | Baseline(Day0), Day 14, Day 28 and Day 56
Change in Lissamine Green Conjunctival Staining(LGCS) score from baseline to Day 14, Day 28, Day 56 and Day 84 | Baseline(Day0), Day 14, Day 28, Day 56 and Day 84
Change in Schirmer Test score from baseline to Day 14, Day 28, Day 56 and Day 84 | Baseline(Day0), Day 14, Day 28, Day 56 and Day 84
Change in Tear Break-Up Time(TBUT) from baseline to Day 14, Day 28, Day 56 and Day 84 | Baseline(Day0), Day 14, Day 28, Day 56 and Day 84
Change in Standard Patient Evaluation of Eye Dryness questionnaire(SPEED) from baseline to Day 14, Day 28, Day 56 and Day 84 | Baseline(Day0), Day 14, Day 28, Day 56 and Day 84
Total number of artificial tears use during the 12 weeks of treatment period | Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Choun-Ki Joo, M.D.,Ph.D., Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No